CLINICAL TRIAL: NCT00329043
Title: A Phase II Neoadjuvant Trial of Sunitinib Malate (SU011248) Plus Hormonal Ablation for Patients Who Have High Risk Localized Prostate Cancer and Will Undergo Prostatectomy
Brief Title: Sunitinib Malate With Hormonal Ablation for Patients Who Will Have Prostatectomy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0903; NCI-2012-01364 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-05-19; First posted 2006-05-24 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Adenocarcinoma of the Prostate; Ductal Adenocarcinoma of the Prostate; Hormonal Ablation; Radical Prostatectomy; LHRH Agonist; Lupron; Leuprolide; Sunitinib Malate; SU011248
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sunitinib + Hormonal Ablation Before Prostatectomy (Experimental): Sunitinib Malate 25 to 37.5 mg/day once daily for 30 days (= 1 cycle), up to 3 cycles. LHRH Agonist intramuscular injection either monthly for 3 months or in a single 3-month dose. Radical prostatectomy after completion of Sunitinib and LHRH agonist.
  Interventions: Drug: LHRH Agonist; Drug: Sunitinib Malate; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: LHRH Agonist — Intramuscular injection either monthly for 3 months or in a single 3-month dose.
  Other Names: Lupron; Leuprolide
Drug: Sunitinib Malate — 25 to 37.5 mg/day once daily for 30 days (= 1 cycle), up to 3 cycles.
  Other Names: SU011248
Procedure: Radical Prostatectomy — Radical prostatectomy after completion of Sunitinib and LHRH agonist.

SUMMARY:
The goal of this clinical research study is to learn if the addition of sunitinib malate (SU011248) to hormone based castration is an effective treatment for shrinking or controlling the tumor before having the prostate removed.

DETAILED DESCRIPTION:
Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer. Hormonal treatment is used to lower testosterone levels in the body because prostate cancer cells need testosterone to survive.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your complete medical history will be recorded. You will have a physical exam, including measurement of vital signs (blood pressure, pulse, temperature, and weight). Blood (about 2 teaspoons) and urine will be collected for routine tests. You will have a computerized tomography (CT) or magnetic resonance imaging (MRI) scan, a bone scan, or a chest x-ray to evaluate the status of your disease. You will be asked about any medications or treatments you are currently taking. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart) and an echocardiogram. An echocardiogram uses sound waves to make pictures of your heart, which helps show how well your heart pumps blood. You will be asked to lie on your left side while a technician places a probe with gel on your chest to create images of your heart to determine the function and size. Your ability to perform daily activities will also be evaluated. You will have a bone marrow aspirate and biopsy. To collect a bone marrow aspirate and biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

If you are found to be eligible to take part in this study, you will take the sunitinib malate by mouth 1 time a day for 30 days together with hormonal ablation therapy. You will receive hormone injections to lower the levels of testosterone in the blood. Hormonal therapy may be given either monthly for 3 months or in a single 3-month dose. Every 30 days is considered a study "cycle." You may receive up to 3 cycles of treatment.

On Day 1 of each cycle, you will have a physical exam and you will be asked about your medical history. Blood (about 2 teaspoons) will be drawn for routine tests. You will be asked about any medications you have taken and any side effects you may have experienced. You will be asked questions about your ability to perform daily activities (performance status evaluation.)

On Day 15 of Cycle 1, you will be asked about any side effects you have experienced. Blood (about 2 teaspoons) will be drawn for routine testing.

After completing 3 cycles of treatment, you will have surgery to remove your prostate. The surgery will occur 1-2 weeks after you receive the last dose of study drug.

After the last dose of the study drug, you will have a follow-up visit. You will be asked about any side effects you are experiencing and you will have a physical exam. You will also have digital rectal exam. Blood (about 2 teaspoons) will be drawn for routine tests. You will also have an echocardiogram. An echocardiogram uses sound waves to make pictures of your heart, which helps show how well your heart pumps blood. You will be asked to lie on your left side while a technician places a probe with gel on your chest to create images of your heart to determine the function and size.

You will have a follow-up visit, 28 days after you stop treatment. You will have a physical exam and your complete medical history will be recorded. Blood (about 2 teaspoons) will be drawn for routine tests. You will be asked about any medications you have taken and any side effects you may have experienced. You will have a performance status evaluation. You will have an echocardiogram if it was abnormal at your last visit.

About 3 months after your surgery, you will return for another follow-up visit. You will have a physical exam and your complete medical history will be recorded. Blood (about 2 teaspoons) will be drawn for routine tests. You will have a performance status evaluation.

For the first year after surgery you will have a prostate specific antigen (PSA) blood test every 3 months. Two (2) years after surgery you will begin having PSA tests every 6 months.

This is an investigational study. Sunitinib malate has been authorized by the FDA for research purposes only. About 64 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed adenocarcinoma of the prostate that in the opinion of the surgeon is resectable. Ductal adenocarcinoma of the prostate is included.
2. All patients must be regarded as low anesthetic risk for radical prostatectomy and confirm their intention to undergo radical prostatectomy at the end of the neoadjuvant therapy.
3. All patients must have one of the following high-risk features: clinical (c) T(subscript)3 disease or Gleason 8-10 adenocarcinoma or cT(subscript)2(subscript)b-c and PSA >= 10 ng/ml and Gleason 7 adenocarcinoma. The 1992 AJCC staging system will be followed.
4. ECOG performance status 0 or 1.
5. Prior hormonal therapy up to 2 months is permitted.
6. Patients must have adequate bone marrow function defined as an absolute peripheral granulocyte count of >= 1,500/mm^3 and platelet count of >= 100,000/mm^3; hemoglobin >= 9.0g/dl; adequate hepatic function defined as a total bilirubin of <=1.5 mg/dl and AST/ALT <= 2 x the upper limit of normal; adequate renal function defined as serum creatinine <= 1.5 x the upper limits of normal or creatinine clearance >= 40cc/min (measured or calculated).
7. Patients must sign the current IRB approved informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution.
8. All patients must have a surgical and medical oncology consult prior to signing informed consent.

Exclusion Criteria:

1. Patients with small cell or sarcomatoid prostate cancers are not eligible.
2. Patients with clinical or radiological evidence of metastatic disease.
3. Patients receiving ketoconazole as a prior hormonal therapy.
4. Prior chemotherapy or experimental agents for prostate cancer.
5. Patients with any infection process, in the criterion of the investigator, that could worsen or its outcome be affected, as a result of the investigational therapy.
6. Patients with NYHA Class III/IV congestive heart failure, unstable angina, cerebrovascular accident or transient ischemic attack, or pulmonary embolism or myocardial infarction in the last 6 months.
7. Uncontrolled severe hypertension (>= 140/90 despite controlling medication), uncontrolled diabetes mellitus, oxygen-dependent lung disease, known chronic liver disease or HIV infection.
8. Second malignancies (excluding non-melanoma skin cancer) unless disease-free for 3 years.
9. Ongoing treatment with therapeutic doses of coumadin. However, low dose coumadin up to 2mg PO daily for deep vein thrombosis prophylaxis is allowed. Low molecular weight heparin is allowed.
10. Overt psychosis, mental disability or otherwise incompetent to give informed consent or history of non-compliance.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2006-05-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Pathological Complete Response (pCR) | Surgery following 3 months of therapy.
  Response defined as pathological complete remission based on operative findings and tissue obtained at surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org